CLINICAL TRIAL: NCT00499954
Title: An Open, Mono-Centre Trial to Investigate the Correlation Between Concentrations of Glucose in Arterialized Venous Blood and Subcutaneous Interstitial Fluid Applying Different Extracorporeal Sensor Techniques in Type 1 Diabetics
Brief Title: Investigation of Correlation Between Concentrations of Glucose in Blood and Interstitial Fluid in Type 1 Diabetics
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Other Study IDs: CM9 diabetes_sensor
Record Dates: First submitted 2007-07-11; First posted 2007-07-12 (Estimated); Last update posted 2007-07-12 (Estimated); Status verified 2006-04

CONDITIONS: Type 1 Diabetes
Keywords: microdialysis; subcutaneous adipose tissue; glucose sensor; glucose monitoring; type 1 diabetes; Guardian RT; Glucoday S
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Microdialysis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Microdialysis
Device: Guardian RT
Device: Glucoday S

SUMMARY:
This is a mono-centre trial performed at the Center for Clinical Research at the Medical University Graz. There will be a screening information and a study visit.In the study visit arterialized venous blood glucose values will be monitored and subcutaneous sampling of interstitial fluid (ISF) with microdialysis for glucose determination will be performed. Additionally to the laboratory analysis of the subcutaneous glucose samples, the glucose will be measured with extracorporeal on-line sensors and two marketed devices (Guardian RT and Glucoday S).The study visit will last 30 hours starting with the insertion of microdialysis catheters in the abdominal subcutaneous tissue and the insertion of the catheters for the Glucoday S system and Guardian RT system. The primary hypothesis of the study is: Interstitial fluid glucose concentration profiles correlate to the arterialized venous blood glucose concentration profile in type 1 diabetic subjects.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained before any trial-related activities.
* Skin fold thickness of minimally 5 mm
* Age of patients in the range from 19 to 60 years.
* Type 1 diabetes

Exclusion Criteria:

* Severe acute and/or chronic diseases
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or co-operation.
* Taking of any vasoactive substances or anticoagulation medication.
* Diseases of the skin which could interfere with application of the catheters
* Pregnancy or breastfeeding

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2006-02

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Pieber, MD, Principal Investigator — Medical University Graz, Graz, Austria
Locations (1):
- Medical University Graz - Clinical Research Center, Graz, Styria, Austria